CLINICAL TRIAL: NCT01129102
Title: Phase 3, Placebo Controlled, Randomized, Double-blinded, Nonsteroidal Antiinflammatory Drug add-on, Clinical Trial of NPC-01 for Treatment of Dysmenorrhea
Brief Title: Efficacy and Safety Study of NPC-01 to Treat Dysmenorrhea
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Nobelpharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NPC-01-2
Record Dates: First submitted 2010-05-21; First posted 2010-05-24 (Estimated); Results first posted 2014-06-17 (Estimated); Last update posted 2025-03-05 (Actual); Status verified 2025-02

CONDITIONS: Dysmenorrhea
MeSH Terms: conditions — Dysmenorrhea

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- NPC-01 (Experimental): Norethisterone 1mg, Ethinyl estradiol 0.02mg
  Interventions: Drug: NPC-01
- IKH-01 (Active Comparator): Norethisterone 1mg, Ethinyl estradiol 0.035mg
  Interventions: Drug: IKH-01
- Placebo (Placebo Comparator): Placebo for NPC-01
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NPC-01 — Norethisterone 1mg, Ethinyl estradiol 0.02mg
  Arms: NPC-01
Drug: IKH-01 — Norethisterone 1mg, Ethinyl estradiol 0.035mg
  Arms: IKH-01
Drug: Placebo — Placebo for NPC-01
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether NPC-01 is effective in the treatment of dysmenorrhea.

DETAILED DESCRIPTION:
The main objective of this study is to confirm the effectiveness and safety profile of NPC-01 in comparison with placebo in the treatment of dysmenorrhea (primary and secondary dysmenorrhea).

Additionally we also investigate the differences of effectiveness of NPC-01 in comparison with IKH-01 in the treatment of secondary dysmenorrhea as a reference, because IKH-01 is already marketed at them.

To achieve these, closed testing procedure is used in this study. After confirming statistical differences between NPC-01 and Placebo in the total dysmenorrhea, stratified analysis is carried out for primary dysmenorrhea (NPC-01, Placebo), and secondary dysmenorrhea (NPC-01, IKH-01 and Placebo).

ELIGIBILITY:
Inclusion Criteria:

* dysmenorrhea

Exclusion Criteria:

* severe hepatopathy
* pregnant woman

Min Age: 16 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 215 (Actual)
Dates: Start 2010-05; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Naoki Terakawa, M.D.,Ph.D., Study Director — Nissay Hospital,Osaka,Japan

REFERENCES:
- [Derived] Schroll JB, Black AY, Farquhar C, Chen I. Combined oral contraceptive pill for primary dysmenorrhoea. Cochrane Database Syst Rev. 2023 Jul 31;7(7):CD002120. doi: 10.1002/14651858.CD002120.pub4. PMID 37523477
- [Derived] Harada T, Momoeda M. Evaluation of an ultra-low-dose oral contraceptive for dysmenorrhea: a placebo-controlled, double-blind, randomized trial. Fertil Steril. 2016 Dec;106(7):1807-1814. doi: 10.1016/j.fertnstert.2016.08.051. Epub 2016 Oct 4. PMID 27717552

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | NPC-01 | IKH-01 | Placebo
Started | 110 | 50 | 55
Completed | 102 | 44 | 48
Not Completed | 8 | 6 | 7
Not completed — No study drug treatment | 2 | 3 | 1
Not completed — Withdrawal by Subject | 2 | 0 | 3
Not completed — Protocol Violation | 0 | 1 | 1
Not completed — Pregnancy | 0 | 0 | 1
Not completed — Adverse Event | 2 | 2 | 1
Not completed — Lost to Follow-up | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline analysis population was carried out based on FAS data set. 110, 50 and 55 pts were assigned to NPC-01, IKH-01 and placebo, respectively, and administered study drug 108, 47 and 54 pts. Safety and FAS analysis was carried out on 107, 47 and 54 pts/105, 47 and 54 pts due to 1 and 2 pts of NPC-01 have no available data respectively.
Groups:
- Total: Total of all reporting groups
Arm/Group | NPC-01 | IKH-01 | Placebo | Total
Number analyzed (Participants) | 105 | 47 | 54 | 206
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.4 (7.29) | 34.0 (6.93) | 30.4 (7.41) | 32.3 (7.21)
Age, Customized [Number; unit: participants]
  Under 30 years of age | 39 | 13 | 29 | 81
  30 year of age and older | 66 | 34 | 25 | 125
Sex/Gender, Customized [Number; unit: participants]
  Female | 105 | 47 | 54 | 206
Diagnostic categories [Number; unit: participants]
  Primary dysmenorrhea | 55 | 0 | 28 | 83
  Secondary dysmenorrhea | 50 | 47 | 26 | 123
Total dysmenorrhea score [Mean (Standard Deviation); unit: units on a scale] — The detail of dysmenorrhea score that was used in this study is the following. These subscales summed for a total dysmenorrhea score (minimum 0 to maximum 6). Pain score None 0 : None Mild 1 : There are some troubles for work Moderate 2 : Needing to rest in bed and/or affecting work Severe 3 : Morre than 1 day in bed and not possible to work
  Drug score (during a menstrual period) None 0 : None Mild 1 : taking analgesics for 1 days Moderate 2 : taking analgesics for 2 days Severe 3 : taking analgesics more than 3 days
  units on a scale
    Total dysmenorrhea | 4.1 (1.00) | NA (NA) — IKH-01 was not allocated for primary dysmenorrhea in this study. Therefore, total dysmenorrhea score is not available for IKH-01 group. | 4.2 (0.95) | NA (NA) — Data unavailable for IKH-01 group
    Primary dysmenorrhea | 3.9 (0.92) | NA (NA) — IKH-01 was not allocated for primary dysmenorrhea in this study. | 4.3 (0.90) | NA (NA) — Data unavailable for IKH-01 group
    Secondary dysmenorrhea | 4.3 (1.05) | 4.0 (0.87) | 4.1 (0.99) | 4.1 (0.96)
Visual analogue scale (VAS) for primary dysmenorrhea [Mean (Standard Deviation); unit: units on a scale] — VAS stands for Visual Analogue Scale of pain. The scale was rated as a graphic rating scale. as a 100mm baseline from 0:No pain to 100:Worst possible pain.
  units on a scale | 51.8 (20.57) | NA (NA) — IKH-01 was not allocated for primary dysmenorrhea in this study. Therefore, VAS for primary dysmenorrhea is not available for IKH-01 group. | 48.6 (20.15) | NA (NA) — Data unavailable for IKH-01 group

OUTCOME MEASURES:

1. Primary Outcome: Patient Response to Treatment for Dysmenorrhea, as Evaluated by Difference of Total Dysmenorrhea Score (Baseline/Pretreatment-End of Treatment)
Description: The detail of dysmenorrhea score that was used in this study is the following. These subscales summed for a total dysmenorrhea score (minimum 0 to maximum 6). Pain score None 0 : None Mild 1 : There are some troubles for work Moderate 2 : Needing to rest in bed and/or affecting work Severe 3 : Morre than 1 day in bed and not possible to work
  Drug score (during a menstrual period) None 0 : None Mild 1 : taking analgesics for 1 days Moderate 2 : taking analgesics for 2 days Severe 3 : taking analgesics more than 3 days
Time Frame: 16weeks
Population: Primary endpoints were analysed based on FAS population. Data unavailable for IKH-01 group because IKH-01 group only assigned for secondary dysmenorrhea.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | NPC-01 | Placebo
Number analyzed (Participants) | 105 | 54
units on a scale
  Pretreatment | 4.1 (1.00) | 4.2 (0.95)
  End of treatment | 1.8 (1.57) | 2.9 (1.55)

2. Secondary Outcome: Difference in the VAS of Primary Dysmenorrhea (Baseline/Pretreatment-End of Treatment)
Description: VAS stands for Visual Analogue Scale of pain. The scale was rated as a graphic rating scale. as a 100mm baseline from 0:No pain to 100:Worst possible pain.
Time Frame: 16weeks
Population: This analysis was carried out based on FAS population. IKH-01 was not allocated for primary dysmenorrhea in this study. Therefore, VAS for primary dysmenorrhea is not available in IKH-01 group.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | NPC-01 | Placebo
Number analyzed (Participants) | 105 | 54
units on a scale
  Pretreatment | 51.8 (20.57) | 48.6 (20.15)
  End of treatment | 21.2 (20.18) | 35.6 (21.74)

ADVERSE EVENTS:
Time Frame: From initiation of study drug to end of 6 cycle of menstrual, an average of 6 months
Arm/Group | NPC-01 | IKH-01 | Placebo
Serious Adverse Events (participants affected / at risk) | 0/107 | 1/47 | 0/54
Other Adverse Events (participants affected / at risk) | 103/107 | 45/47 | 44/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NPC-01 (N=107) | IKH-01 (N=47) | Placebo (N=54)
Abdominal pain lower (Dysmenorrhoea aggravated) (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NPC-01 (N=107) | IKH-01 (N=47) | Placebo (N=54)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (2) | 3 (4)
Abdominal pain (Gastrointestinal disorders) | 6 (9) | 1 (1) | 1 (1)
Abdominal pain lower (Gastrointestinal disorders) | 12 (19) | 2 (3) | 1 (3)
Abdominal pain upper (Gastrointestinal disorders) | 5 (5) | 3 (4) | 4 (4)
Nausea (Gastrointestinal disorders) | 13 (17) | 10 (12) | 3 (5)
Vomiting (Gastrointestinal disorders) | 3 (3) | 3 (3) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 3 (3) | 2 (3)
Gastroenteritis (Infections and infestations) | 5 (5) | 2 (2) | 3 (3)
Nasopharyngitis (Infections and infestations) | 42 (71) | 12 (16) | 19 (31)
Vulvovaginal candidiasis (Infections and infestations) | 0 (0) | 1 (1) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 3 (3)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3) | 0 (0)
Headache (Nervous system disorders) | 25 (41) | 10 (17) | 4 (6)
Hypomenorrhoea (Reproductive system and breast disorders) | 7 (7) | 1 (1) | 0 (0)
Menorrhagia (Reproductive system and breast disorders) | 6 (7) | 5 (5) | 0 (0)
Metrorrhagia (Reproductive system and breast disorders) | 75 (165) | 37 (71) | 21 (35)
Oligomenorrhoea (Reproductive system and breast disorders) | 30 (38) | 7 (9) | 9 (10)
Polymenorrhoea (Reproductive system and breast disorders) | 9 (12) | 5 (5) | 0 (0)
Breast discomfort (Reproductive system and breast disorders) | 8 (10) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
There is an agreement between the sponsor and PI that no restricts the PI's right but need to discuss the timing of publish date of trial results after the trial is completed.